CLINICAL TRIAL: NCT05552534
Title: Impact of an Intervention of Screening, Treatment Initiation and Referral to Promote Smoking Cessation in Emergency Department Patients: the Pilot PROSCEED Randomized Controlled Study
Brief Title: Impact of an Intervention of Screening, Treatment Initiation and Referral to PROmote Smoking CEssation in Emergency Department Patients
Acronym: PROSCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220066; ID RCB 2021-A03003-38 (Other: ANSM)
Record Dates: First submitted 2022-04-04; First posted 2022-09-23 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Cessation
Keywords: Emergency medicine; Public Health; Addictionology; Smoking cessation; Tobacco dependence treatment
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: STIR PROTOCOL
- Control group (No Intervention)

INTERVENTIONS:
Other: STIR PROTOCOL — Screening, STIR protocol (screening, brief intervention, incentive to download the tobacco info service application, delivery of the "tobacco-info-service" brochure, initiation of a nicotine patch made by the trained emergency nurse or doctor) then three consultations face-to-face or remotely with a member of the team addictionology at 7 days, 1 and 3 months.
  Arms: Intervention group

SUMMARY:
Smoking cessation assistance is one of the major issues in prevention policies because the prevalence of smoking remains high in France. With its numerous consultations, an emergency service seems to be an interesting place for setting up and helping with weaning, despite specific working conditions. The study, which is a pilot, is interested in the feasibility and efficacy of the implementation of a STIR (Screening, Treatment Intervention and Referral) protocol, which screening, brief intervention, nicotine replacement therapy and referral to a specialist in order to help the patients in smoking cessation.

DETAILED DESCRIPTION:
Individual randomization as soon as the patient gives his consent and meets the inclusion - non-inclusion criteria.

Control group: delivery of the "tobacco-info-service" brochure titled "Why quit smoking? ", then phone call at 7 days and a month to collect tobacco consumption. Visit for 3 month. Intervention group: STIR protocol (screening, brief intervention, incentive to download the tobacco info service application, delivery of the "tobacco-info-service" brochure, initiation of a nicotine replacement therapy with nicotine patches made by a trained emergency nurse or doctor, then three consultations face-to-face or remotely with a member of the team addictionology at 7 days, 1 and 3 months.

In both groups: collection of the primary endpoint during the M3 visit. For patients who did not come (regardless of the group):

call for collection of the main judgment criterion

Carers will be included and will sign a consent form once the eligibility criteria have been checked and consent has been signed. They will be asked to complete an adherence questionnaire (Likert scale) regarding smoking prevention in emergency departments before the start of the study and after the last patient follow-up has taken place.

ELIGIBILITY:
Inclusion Criteria:

* Age >= to 18 years old
* Active smoker defined by having smoked at least 100 cigarettes in total in his life, associated with daily consumption or weekly
* Free and informed consent signed by the patient
* Patient with an understanding of the French language to participate in the intervention if necessary
* Patient affiliated to a social security regimen

Care giver inclusion criteria:

* Age ≥ 18 years
* Caregiver working in one of the 3 departments participating in the study
* Signature of free and informed consent

Exclusion Criteria:

* Absolute vital emergency
* Pregnant or breastfeeding women
* Contraindication to taking nicotine
* Taking nicotine by patch or gum or e-cigarette
* Patient under AME (national medical insurance)
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Feasibility and efficacy of a smoking cessation intervention | 3 months after emergency consultation
  Composite outcome: Proportion of patients who participated in follow-up consultations at 3 months after going to the emergency room and proportion of patients weaned from smoking at three months in the intervention group, compared to the control group.
  A patient is said to be weaned if he / she declares having stopped smoking for 7 days 3 months after his / her visit to the emergency room

SECONDARY OUTCOMES:
proportion of patients who participated in consultations at D7 and M1 | Day 7 and 1 month after emergency consultation
  Assessment of the patient circuit
description of the procedure (duration of the inclusion) | 4 months
  Description of the research circuit
number of patients who refused to participate | 4 months
  Description of the procedure's barriers
Number of doctors/paramedics involved, and of staff who performed the follow-up | 4 months
  Description of staff involved
Feasibility of measuring exhaled carbon monoxide | 3 months after emergency consultation
  Proportion of patients with a carbon monoxide measurement expired
Correlation of the measurement of exhaled carbon monoxide and declaration of withdrawal | 3 months after emergency consultation
Effectiveness of the smoking cessation intervention | Day 7 and 1 month after emergency consultation
  Proportion of patients weaned at 7 days and at 1 month assessed, declarative, collected by phone
Number of smoked cigarettes | Day 7, 1 month and 3 month after emergency consultation
  Number of cigarettes smoked daily at 7 days, 1 and 3 months, declarative
Patients' adherence to the intervention | 3 month after emergency consultation
  - Questionnaire with Likert scale: In order to measure adherence to the intervention, 13 sentences in favor of the intervention : answers from 1. I strongly disagree to 5 . I completely agree.
  A higher score mean a better adherence (min: 13, max : 65).
  - Proportion of patients who completed follow-up consultations at 7 days and one month
Emergency teams' adherence to the intervention | 3 month after emergency consultation
  Questionnaire with Likert scale: In order to measure adherence to the intervention, 11 sentences in favor of the intervention : answers from 1. I strongly disagree to 5 . I completely agree.
  A higher score mean a better adherence (min: 11, max : 55).
Patients ' adherence to the intervention, according to demographic criteria. | 3 month after emergency
  Description of the population according to age, gender, socio-economic characteristics, grounds for appeal

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laure Philippon, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No